CLINICAL TRIAL: NCT06584539
Title: Online Randomized Experiment Evaluating Eco-Labels on Restaurant Menus
Brief Title: Eco-labels on Restaurant Menus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Joshua Petimar, Assistant Professor, Population Medicine, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000970
Record Dates: First submitted 2024-08-09; First posted 2024-09-05 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Nutrition; Food Selection; Food Preferences; Dietary Habits; Healthy Diet
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eco-labels (Experimental): Participants will view a mock restaurant menu based on a popular US sit-down restaurant. They will be instructed to select the item or items they would like to order from the restaurant. The menu will display eco-labels next to more sustainable menu appetizers and entrees (i.e., appetizers and entrees that are in the bottom half of carbon footprints [i.e., greenhouse gas emissions in CO2-equivalents associated with production of the item] among appetizers and entrees).
  Interventions: Behavioral: Eco-Labels
- Control (No Intervention): Participants will view a mock restaurant menu based on a popular US sit-down restaurant. They will be instructed to select the item or items they would like to order from the restaurant. The menus will not display eco-labels.

INTERVENTIONS:
Behavioral: Eco-Labels — Eco-labels will be displayed next to more sustainable restaurant menu items. The labels will display an earth icon and the words "ENVIRONMENTALLY FRIENDLY."
  Arms: Eco-labels

SUMMARY:
The goal of this study is to determine whether eco-labels denoting more sustainable menu items improve the healthfulness of participants' entrée and appetizer selections from a restaurant menu. US adults will complete a restaurant ordering task in which they will select menu items to order from a mock restaurant menu modeled after a popular US sit-down restaurant. Participants will be randomized to a restaurant menu with or without eco-labels denoting more sustainable menu items. The investigators will record participants' selections from the menu. Participants will also answer survey questions.

DETAILED DESCRIPTION:
The goal of this study is to determine whether eco-labels denoting more sustainable menu items improve the healthfulness of participants' entrée and appetizer selections. The survey research company Cloud Research will recruit a sample of approximately 3,100 US adults ages 18+ who read and speak English.

Participants will complete a between-subjects online randomized experiment. They will perform a restaurant ordering task in which they will select menu items to order from a mock restaurant menu modeled after a popular US sit-down restaurant. They will be randomized to 1 of 2 conditions: 1) eco-labels or 2) control. In the eco-labels condition, participants will order from a restaurant menu with eco-labels next to more sustainable menu items. In the control condition, participants will order from a restaurant menu without eco-labels. The investigators will record participants' selections from the menu. After completing the ordering task, participants will complete an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Reside in the US
* Can read and speak English

Exclusion Criteria:

* Under the age of 18 years
* Reside outside of the United States
* Unable to complete a survey in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3147 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Healthfulness of participants' entrée and appetizer selections | Through study completion, an average of 15 minutes
  The study will assess the healthfulness of participants' entrée and appetizer selections as the average Ofcom Nutrient Profiling Model score of the entrees and appetizers the participants select in the restaurant ordering task. Ofcom Nutrient Profiling Model scores will be calculated for each item participants select. Items receive higher Ofcom scores when they contain lower calorie, saturated fat, sodium, and sugar density, higher protein and fiber density, and more fruits, vegetables, legumes, and nuts. The investigators will calculate the average score across participants' entrée and appetizer selections. The Ofcom Nutrient Profiling Model score ranges from 0 to 100, where higher scores indicate healthier products.

SECONDARY OUTCOMES:
Healthfulness of participants' restaurant selections | Through study completion, an average of 15 minutes
  The study will assess the healthfulness of participants' restaurant selections as the average Ofcom Nutrient Profiling Model score of the menu items the participants select in the restaurant ordering task. Ofcom Nutrient Profiling Model scores will be calculated for each item participants select. Items receive higher Ofcom scores when they contain lower calorie, saturated fat, sodium, and sugar density, higher protein and fiber density, and more fruits, vegetables, legumes, and nuts. The investigators will calculate the average score across participants' selections. The Ofcom Nutrient Profiling Model score ranges from 0 to 100, where higher scores indicate healthier products.
Calories selected from all items | Through study completion, an average of 15 minutes
  The study will assess the number of calories participants select in the restaurant ordering task, calculated as the total number of calories selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher calories selected.
Calories selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the number of calories participants select from entrees and appetizers in the restaurant ordering task, calculated as the total number of calories selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher calories selected.
Sodium selected from all items | Through study completion, an average of 15 minutes
  The study will assess the amount of sodium participants select in the restaurant ordering task, calculated as the total sodium (in milligrams) selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher sodium selected.
Sodium selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the amount of sodium participants select from entrees and appetizers in the restaurant ordering task, calculated as the total sodium (in milligrams) selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher sodium selected.
Saturated fat selected from all items | Through study completion, an average of 15 minutes
  The study will assess the amount of saturated fat participants select in the restaurant ordering task, calculated as the total saturated fat (in grams) selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher saturated fat selected.
Saturated fat selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the amount of saturated fat participants select from entrees and appetizers in the restaurant ordering task, calculated as the total saturated fat (in grams) selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher saturated fat selected.
Sugar selected from all items | Through study completion, an average of 15 minutes
  The study will assess the amount of sugar participants select in the restaurant ordering task, calculated as the total sugar (in grams) selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher sugar selected.
Sugar selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the amount of sugar participants select from entrees and appetizers in the restaurant ordering task, calculated as the total sugar (in grams) selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher sugar selected.
Fiber selected from all items | Through study completion, an average of 15 minutes
  The study will assess the amount of fiber participants select in the restaurant ordering task, calculated as the total fiber (in grams) selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher fiber selected.
Fiber selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the amount of fiber participants select from entrees and appetizers in the restaurant ordering task, calculated as the total fiber (in grams) selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher fiber selected.
Protein selected from all items | Through study completion, an average of 15 minutes
  The study will assess the amount of protein participants select in the restaurant ordering task, calculated as the total protein (in grams) selected across all menu items the participant selected in the restaurant ordering task. Higher values indicate higher protein selected.
Protein selected from entrees and appetizers | Through study completion, an average of 15 minutes
  The study will assess the amount of protein participants select from entrees and appetizers in the restaurant ordering task, calculated as the total protein (in grams) selected across entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate higher protein selected.
Carbon footprint of all items selected | Through study completion, an average of 15 minutes
  The study will assess the carbon footprint of all items that participants select in the restaurant ordering task, calculated as the total carbon footprint (in CO2-equivalents) selected across all items the participant selected in the restaurant ordering task. Higher values indicate a larger carbon footprint of selected items.
Carbon footprint of entrees and appetizers selected | Through study completion, an average of 15 minutes
  The study will assess the carbon footprint of all entrees and appetizers that participants select in the restaurant ordering task, calculated as the total carbon footprint (in CO2-equivalents) selected across all entrees and appetizers the participant selected in the restaurant ordering task. Higher values indicate a larger carbon footprint of selected items.
Noticing of eco-labels | Through study completion, an average of 15 minutes
  The study will assess noticing of the eco-labels with 1 item: "When you were selecting items to order, did you notice any other labels next to menu items?" Response options will be "yes" (coded as 1) and "no" (coded as 0).
Thinking about the environmental effects of food | Through study completion, an average of 15 minutes
  The study will assess thinking about the environmental effects of food while ordering with 1 item: "When you chose what to order from the menu, how much did you think about each of the following characteristics? Environmental sustainability." Response options will range from "Not at all" (coded as 1) to "A great deal" (coded as 5). Higher scores indicate more thinking about the environmental effects of food while ordering.
Thinking about the healthfulness of food | Through study completion, an average of 15 minutes
  The study will assess thinking about the healthfulness of food while ordering with 1 item: "When you chose what to order from the menu, how much did you think about each of the following characteristics? Healthfulness." Response options will range from "Not at all" (coded as 1) to "A great deal" (coded as 5). Higher scores indicate more thinking about the healthfulness of food while ordering.
Thinking about the taste of food | Through study completion, an average of 15 minutes
  The study will assess thinking about the taste of food while ordering with 1 item: "When you chose what to order from the menu, how much did you think about each of the following characteristics? Taste." Response options will range from "Not at all" (coded as 1) to "A great deal" (coded as 5). Higher scores indicate more thinking about the taste food while ordering.
Perceived sustainability of sustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived sustainability of sustainable menu items with 1 item: "How environmentally sustainable do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 more sustainable menu items. For participants in the ecolabels arm, the item will display an ecolabel. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived sustainability.
Perceived healthfulness of sustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived healthfulness of sustainable menu items with 1 item: "How healthy do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 more sustainable menu items. For participants in the ecolabels arm, the item will display an ecolabel. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived healthfulness.
Perceived tastiness of sustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived tastiness of sustainable menu items with 1 item: "How tasty do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 more sustainable menu items. For participants in the ecolabels arm, the item will display an ecolabel. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived tastiness.
Perceived sustainability of unsustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived sustainability of unsustainable menu items with 1 item: "How environmentally sustainable do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 less sustainable menu items. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived sustainability.
Perceived healthfulness of unsustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived healthfulness of unsustainable menu items with 1 item: "How healthy do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 less sustainable menu items. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived healthfulness.
Perceived tastiness of unsustainable menu items | Through study completion, an average of 15 minutes
  The study will assess perceived tastiness of unsustainable menu items with 1 item: "How tasty do you think this item is?" For this question, participants will be randomized to view an image of 1 of 13 less sustainable menu items. Response options will range from "Not at all" (coded as 1) to "Extremely" (coded as 5). Higher scores indicate higher perceived tastiness.

OTHER OUTCOMES:
Liking of the eco-label | Through study completion, an average of 15 minutes
  The study will assess the extent to which participants like the eco-label with 1 item: "I like this label." Response options will range from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5). The investigators will dichotomize responses into agree (4 or 5, indicating participants like the ecolabel) vs. disagree or neutral (1-3, indicating participants do not like the ecolabel).
Wanting to see the eco-label on restaurant menus | Through study completion, an average of 15 minutes
  The study will assess the extent to which participants want to see the eco-label on restaurant menus with 1 item: "I want to see this label on menus next to foods that are more environmentally sustainable." Response options will range from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5). The investigators will dichotomize responses into agree (4 or 5, indicating participants want to see the label on restaurant menus) vs. disagree or neutral (1-3, indicating participants do not want to see the label on restaurant menus).
Label helpfulness in choosing more environmentally sustainable foods | Through study completion, an average of 15 minutes
  The study will assess the extent to which participants think the ecolabel helps them choose more sustainable foods with 1 item: "This label would help me choose more environmentally sustainable foods." Response options will range from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5). The investigators will dichotomize responses into agree (4 or 5, indicating participants think the ecolabel helps them choose more sustainable foods) vs. disagree or neutral (1-3, indicating participants do not think the ecolabel helps them choose more sustainable foods).
Perceptions of control over making sustainable eating decisions | Through study completion, an average of 15 minutes
  The study will assess the extent to which participants perceive that the ecolabel makes them feel more in control of making sustainable eating decisions with 1 item: "This label makes me feel more in control of making sustainable eating decisions." Response options will range from "Strongly disagree" (coded as 1) to "Strongly agree" (coded as 5). The investigators will dichotomize responses into agree (4 or 5, indicating participants perceive the ecolabel increases control over making sustainable eating decisions) vs. disagree or neutral (1-3, indicating participants do not perceive that the ecolabel increases control).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Petimar, ScD, Principal Investigator — Harvard Pilgrim Health Care Institute; Anna Grummon, PhD, Principal Investigator — Stanford University
Locations (1):
- Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will post de-identified individual participant data in a public repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post IDP within 6 months of publication of manuscripts associated with the data generated in this study.
Access Criteria: Data and code will be made publicly available.

REFERENCES:
- [Derived] Grummon AH, Zeitlin AB, Lee CJY, Collis C, Cleveland LP, Musicus AA, Petimar J. Ecolabels and the Healthfulness and Carbon Footprint of Restaurant Meal Selections: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2524773. doi: 10.1001/jamanetworkopen.2025.24773. PMID 40758354

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT06584539/SAP_000.pdf